CLINICAL TRIAL: NCT05179148
Title: Motivational Interviewing for Physical Activity Among Older Adults
Brief Title: MI for Physical Activity Among Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Olayinka Akinrolie, Principal Investigator, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS25249 (H2021:396)
Record Dates: First submitted 2021-12-06; First posted 2022-01-05 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Motivational Interviewing
Keywords: motivational interviewing; physical activity; older adults; virtual
MeSH Terms: conditions — Motor Activity | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Experimental): The arm will receive motivational interviewing
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Motivational Interviewing — MI is a client-centered counselling style for strengthening a person's own motivation and commitment to change. MI helps evoke the person's own motivation for changes through reflective listening, engaging, evoking, and planning

SUMMARY:
The purpose of this study is to determine the feasibility of VIrtual Motivational INTerviewing (VIMINT) to promote physical activity levels among older adults; post-intervention and at two-month follow-up.

DETAILED DESCRIPTION:
Evidence shows that moderate and regular physical activity is associated with the prevention of non-communicable diseases, increased bone density, reduced risk of dementia, and prevention of falls among older adults. Despite the numerous benefits of physical activity, many older adults do not meet the recommended physical activity guidelines of 150 min/week of moderate-to-vigorous intensity physical activity in Canada. MI is a client-centered counselling style for strengthening a person's own motivation and commitment to change. MI helps evoke the person's own motivation for changes through reflective listening, engaging, evoking, and planning. MI has shown to be promising in the general adult population for improving physical activity levels, however, there were mixed results for the effectiveness of MI among older adults. In addition, based on the available evidence, there are no studies evaluating the potential long-term effects of MI on physical activity levels among older adults. This feasibility study is necessary to explore possible challenges that may be encountered in the future larger trial with a two-month follow-up. Due to the recent pandemic (COVID-19), the intervention will be conducted virtually through the videoconferencing platform (Zoom). Therefore, the purpose of this study is to determine the feasibility of VIrtual Motivational INTerviewing (VIMINT) to promote physical activity levels among older adults; post-intervention and at two-month follow-up.

The participants will receive five sessions of the virtual MI over a five-week period through the Zoom platform and each session will last between 45 to 60 minutes. The intervention will be delivered by trained personnel in MI. The MI strategies will include evoking change and guiding participants in establishing goals for improving physical activity. After the 2-month evaluation, counsellors and participants will be invited for a one-on-one Zoom interview. The aim is to explore the perception of the counsellors and participants about the VIMINT study including, views about virtual MI, benefits, and challenges.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 years or older
* living in the community
* able to walk with or without mobility aid for at least 10 metres
* physically inactive i.e., less than 150 minutes of moderate-vigorous intensity
* ready to participate in physical activity and no medical concerns using the Physical Activity Readiness Questionnaire (PAR-Q+)*
* score of ≥ 18 on the telephone version of the Mini-mental State Exam
* able to speak English
* able to have access to a computer, tablet or mobile phone capable of running the videoconferencing platform (Zoom)
* able to access internet and email

Exclusion Criteria:

* • receiving on-going treatment for any medical condition that would prevent safe participation in physical activity

  * living in long-term care
  * participating in other behavioural interventions that focus on improving physical activity

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Total number of participants recruited per month | throughout the study, average of 1 year
  The recruitment rate is the number of participants screened, the number of those who provide written informed consent and the percentage of those who attend the baseline assessment
the percentage of participants that remained after the last data is completed at 1 year | after completion of data collection at 1 year
  Total number of participants that completed the follow-up assessment at 3 months post-baseline divided by the total number of participants that completed the post-intervention assessment at 1 month post-baseline
the counsellor's competence will be assessed using Motivational Interviewing Treatment Integrity Code 4.2.1 after completing the motivational interviewing counselling at 1 month post-baseline assessment | at 1 month post baseline
  The counsellor's competence will be assessed by listening to the audio recorded MI sessions using the global score on the Motivational Interviewing Treatment Integrity Code (MITI 4.2.1.) MITI 4.2.1 consists of four global ratings for the counsellor: cultivating Change talk, Softening Sustain Talk, Partnership, and Empathy. Each of the four global ratings are scored on a five-point Likert scale with "1" and "5" as the lowest and highest proficiency respectively.
participant level of satisfaction will be assessed using the Client Satisfaction Questionnaire version 8 at follow-up assessment which is 3 months post baseline | 3 months post baseline
  The Client Satisfaction Questionnaire version 8 is an 8-item scale that is scored using a Likert from 1 (quite dissatisfied) to 4 (very satisfied). The score ranges from 8 to 32, with a higher score representing higher satisfaction

SECONDARY OUTCOMES:
change from baseline of self-reported light, moderate and vigorous using Community Healthy Activities Model Program for Seniors (CHAMPS) questionnaire at 1 month and 3 months | baseline, 1 month and 3 months post baseline
  CHAMPS is a 41-item questionnaire. We will administer the CHAMPS questionnaire through the Zoom platform at baseline, 1 month, and 3 months post baseline. The participants will be asked to indicate if they engage in an activity, and if the participants indicate "NO" they will be scored zero. Any activities the participants indicate "YES," we will ask how many times they engage in the activity in a week. Afterward, the participants will be asked to select the total hours/week they engage in the activity from the following six categories: less than 1 hr, 1-2½ hrs, 3-4½ hrs, 5-6½ hrs, 7-8½ hrs, and 9 hrs or more. Each activity on the CHAMPS is assigned a Metabolic equivalent (MET) value as recommended by Stewart et al. (2001). We will compute the total hours/week; a MET value of ≥ 3.0 and ≥ 5.0 will be defined as moderate-vigorous and vigorous intensity physical activity respectively.
Change from baseline in the total sporadic minutes per day of the light and moderate-vigorous intensity physical activity and total number of steps per day using activity monitor(GT3X+ model) at 1 months and 3 months | baseline, 1 month and 3 months post baseline
  Participants will be asked to wear the activity monitor on an elastic waistband over the right hip for at least 10 waking hours for seven consecutive days. low frequency extension (LFE) option to capture the various physical activity intensities. The light and moderate-vigorous intensity physical activity will be analyzed using the cut point of 100-759 and ≥760 counts per minute respectively.
Change from baseline in the quality of life using The Research ANd Development-36 (RAND-36) at 1 month and 3 months | baseline, 1month and 3 months post baseline
  RAND-36 is a 36-item generic measure of the HRQoL that assesses eight health concepts: physical functioning (10 items), role limitations due to physical health problem (4 items), role limitations due to emotional problems (3 items), social functioning (2 items), emotional well-being (5 items), energy/fatigue (4 items), pain (2 items), and general health perceptions (5 items). RAND-36 also assesses change in perceived health during the last 12 months using a single item. Each item has different response categories (1-6), which are then transformed to various values as recommended by Hays and Morales (2001). The score ranges between 0 and 100 (SD =10) with a higher score indicating better physical or mental health.
change from baseline in the mean self-efficacy for exercise using 9-item Self-efficacy for exercise questionnaire at 1 month and 3 months | baseline, 1month and 3 months post baseline
  It is a 9-item instrument with responses ranging from 0 (not confident) to 10 (very confident), and a higher score indicating higher self-efficacy for physical activity or exercise. The scoring is calculated by summing up the total score and dividing by the number of items (nine).
change from baseline in the mean of task self-efficacy physical activity using 10 items from task self-efficacy physical activity questionnaire at 1 month and 3 months post baseline. | baseline, 1month and 3 months post baseline
  the self-efficacy physical activity questionnaire is a 10-item, participants will be asked to rate their level of confidence on a scale 0 (not at all confidence) and 100 (completely confident). The ratings will be summed and averaged to give a score of task self-efficacy physical activity score.
change from baseline in the readiness of the participant to change behaviour using readiness-to-change ruler at baseline and 1 month post baseline | baseline and 1 month post baseline
  the readiness-to-change ruler is an arbitrary line on a scale of 0 to 10 where 0 means "Not ready to change," and 10 means "Ready to change''. The readiness-to-change ruler helps to gauge the motivational and ambivalence state of an individual. Typically, the scores are interpreted with 0-3 as "not ready", 4-7 as "ambivalence or not sure" and 8-10 as "ready for change".

CONTACTS AND LOCATIONS:
Overall Officials: Olayinka Akinrolie, MSc, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun F, Norman IJ, While AE. Physical activity in older people: a systematic review. BMC Public Health. 2013 May 6;13:449. doi: 10.1186/1471-2458-13-449. PMID 23648225
- [Background] Vogel T, Brechat PH, Lepretre PM, Kaltenbach G, Berthel M, Lonsdorfer J. Health benefits of physical activity in older patients: a review. Int J Clin Pract. 2009 Feb;63(2):303-20. doi: 10.1111/j.1742-1241.2008.01957.x. PMID 19196369
- [Background] Miller WR, Rollnick S. The methods of motivational interviewing Motivational interviewing: Helping people change. 3rd ed. New York, NY: Guilford press; 2013. p. 29
- [Background] O'Halloran PD, Blackstock F, Shields N, Holland A, Iles R, Kingsley M, Bernhardt J, Lannin N, Morris ME, Taylor NF. Motivational interviewing to increase physical activity in people with chronic health conditions: a systematic review and meta-analysis. Clin Rehabil. 2014 Dec;28(12):1159-71. doi: 10.1177/0269215514536210. Epub 2014 Jun 18. PMID 24942478
- [Background] Brodie DA, Inoue A. Motivational interviewing to promote physical activity for people with chronic heart failure. J Adv Nurs. 2005 Jun;50(5):518-27. doi: 10.1111/j.1365-2648.2005.03422.x. PMID 15882368
- [Background] O'Halloran PD, Shields N, Blackstock F, Wintle E, Taylor NF. Motivational interviewing increases physical activity and self-efficacy in people living in the community after hip fracture: a randomized controlled trial. Clin Rehabil. 2016 Nov;30(11):1108-1119. doi: 10.1177/0269215515617814. Epub 2016 Jul 11. PMID 26603892
- [Background] Quirk F, Dickinson C, Baune B, Leicht A, Golledge J. Pilot trial of motivational interviewing in patients with peripheral artery disease. Int Angiol. 2012 Oct;31(5):468-73. PMID 22990510
- [Background] Akinrolie O, Barclay R, Strachan S, Gupta A, Jasper US, Jumbo SU, et al. The effect of motivational interviewing on physical activity level among older adults: a systematic review and meta-analysis. Physical & occupational therapy In Geriatrics. 2020;38(3):250-63
- See also: Statistic C. Direct measure physical activity of adults, 2012 and 2013 2015 — https://www150.statcan.gc.ca/n1/daily-quotidien/170419/dq170419e-eng.htm